CLINICAL TRIAL: NCT06998381
Title: Ethnic Specificities of S100B Protein Blood Level in Guadeloupe: Cross-sectional Study in Healthy Subjects
Acronym: PS100B-G
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: PAP_RIPH2_2020/18; 2020-A02605-34 (Other: ANSM Frech Human Health Organisation)
Record Dates: First submitted 2025-05-21; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: s100b
Keywords: S100B Protein

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Numerous studies have demonstrated the significant contribution of S100B blood level measurement in the management of minor to moderate traumatic brain injuries, notably by reducing the number of cranial computed tomography (CT) scans by at least one-third. However, physiological blood concentrations of the S100B protein may be higher in individuals with a Black phenotype compared to those with Asian or, in particular, Caucasian phenotypes. Assessing S100B protein levels in healthy individuals will help confirm the variability of its physiological concentration according to skin phenotype.

DETAILED DESCRIPTION:
Thanks to its excellent negative predictive value, the S100B protein has been defined as a reliable alternative to computed tomography (CT) in the management of traumatic brain injury (TBI). Validated by scientific societies in 2014, the use of this biomarker could reduce the number of cerebral CT scans by nearly one-third in cases of minor TBI.

However, implementation of this blood test in routine clinical practice may present challenges. The extrapolation of findings from S100B studies to the context of Guadeloupe remains uncertain. The commonly accepted threshold of 0.1 μg/L for S100B protein, used to determine the need for CT imaging, has been established based on existing literature. Nevertheless, the study by Abdesselam (Clinical Chemistry 49, No. 5, 2003) suggests that S100B concentrations may vary by ethnic background: higher levels have been observed in individuals of Black phenotype (0.14 ± 0.08 μg/L) compared to those of Asian (0.11 ± 0.08 μg/L) and Caucasian (0.07 ± 0.03 μg/L) phenotypes.

A closer analysis of Abdesselam's data reveals that approximately three-quarters of individuals with a Black phenotype may present physiological S100B levels exceeding 0.1 μg/L. Given that the majority of Guadeloupe's population is of Black phenotype, applying the 0.1 μg/L threshold for CT scan decision-making may lack accuracy for this population. Nonetheless, Abdesselam's study involved a limited sample size (46 individuals of Black ethnicity) and showed high interindividual variability in S100B levels. Further validation is therefore required in Guadeloupe and, more broadly, in Caribbean populations.

The planned study will enroll hospital staff who meet predefined eligibility criteria. Prior to inclusion, eligible individuals will receive an information leaflet and consent form, both explained by a physician or a clinical research nurse. Upon obtaining signed informed consent, each subject will complete an anonymous questionnaire detailing ethnic background, age, sex, and weight. A blood sample will then be collected and sent to the biochemistry laboratory at the University Hospital of Guadeloupe for S100B protein analysis.

ELIGIBILITY:
Inclusion Criteria :

* Hospital staff of the University Hospital of Guadeloupe or the Hospital of Basse-Terre
* Age between 18 and 65 years
* Individuals willing to specify their ethnic origin and skin phototype
* Individuals affiliated with or beneficiaries of a social security scheme
* Informed individuals who have given their voluntary, informed, and written consent

Exclusion Criteria :

* Individuals on anticoagulant therapy
* Individuals with a personal history of neurological disease
* Individuals with a personal history of melanoma
* Refusal to participate
* Individuals under guardianship, curatorship, or legal protection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital staff of the University Hospital of Guadeloupe or the Basse-Terre Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
S100B and ethnicity | baseline
  Level of S100B protein expressed in μg / L, which will be compared according to 3 groups: Afro-Caribbean, Indo-Caribbean and Caucasian.

SECONDARY OUTCOMES:
S100B and phototypes | baseline
  Level of S100B protein expressed in μg / L studied according to the 6 phototypes of Fitzpatrick classification.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Delta, MD, Principal Investigator — CHU de la Guadeloupe
Locations (2):
- Guadeloupe (2):
  - CH de la Basse-Terre, Basse-Terre
  - Chu de La Guadeloupe, Pointe-à-Pitre

IPD SHARING:
Plan to Share IPD: Undecided